CLINICAL TRIAL: NCT00733915
Title: A Prospective, Non-Comparative Study to Evaluate the Performance of the DePuy Low Contact Stress (LCS) Complete Mobile-bearing Total Knee System.
Brief Title: Long-term Study of the DePuy Low Contact Stress (LCS) Complete Total Knee System
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT 01/13
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: Arthroplasty, knee, TKA, TKR, Duofix, Porocoat, LCS
MeSH Terms: conditions — Aagenaes syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): Cohort of total knee replacements with LCS Complete knee implants
  Interventions: Device: L.C.S. Complete Knee (DePuy Low Contact Stress Complete Knee System)

INTERVENTIONS:
Device: L.C.S. Complete Knee (DePuy Low Contact Stress Complete Knee System) — L.C.S. Complete mobile-bearing total knee system

SUMMARY:
The main objective of this study is to evaluate how the LCS Complete mobile-bearing total knee system and surgical instrumentation performs.

DETAILED DESCRIPTION:
The secondary objective of this investigation is to evaluate the long-term survivorship and performance of the LCS Complete mobile-bearing total knee system and surgical instrumentation using the American Knee Society Score (AKS) the Oxford Knee Score (OKS), SF-12 and survivorship analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects.
* Subjects who are able to give voluntary, written informed consent to participate in this investigation and from whom consent has been obtained
* Subjects who, in the opinion of the Investigator, are able to understand this investigation, co-operate with the investigational procedures and are willing to return to the hospital for all the required post-operative follow-ups.
* Subjects who present with idiopathic osteoarthritis, rheumatoid arthritis, post traumatic arthritis or any other pathology that in the opinion of the clinical investigator requires a primary total knee arthroplasty and who are considered suitable for treatment with a mobile bearing knee system (LCS Complete).
* Subjects who in the opinion of the Clinical Investigator are considered to be suitable for treatment with the investigation device, according to the indications specified in the package insert leaflet.

Exclusion Criteria:

* Subjects who, in the opinion of the Investigator, have an existing condition that would compromise their participation and follow-up in this study.
* Subjects with a known history of poor compliance to medical treatment.
* Women who are pregnant.
* Subjects who are known drug or alcohol abusers or with psychological disorders that could effect follow-up care or treatment outcomes.
* Subjects involved in Medical-Legal claims.
* Subjects who have participated in a clinical study with an investigational product in the last month.
* Subjects who are currently involved in any injury litigation claims.
* Revision of an existing knee implant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2002-03-01 (Actual); Primary Completion 2007-09-01 (Actual); Study Completion 2014-10-01 (Actual)

PRIMARY OUTCOMES:
To demonstrate the surgical performance of the LCS Complete mobile-bearing total knee system and instrumentation using radiographic and intra-operative assessment | 10 years

SECONDARY OUTCOMES:
To demonstrate the survivorship and performance of the LCS Complete mobile-bearing total knee system using the American Knee Society clinical and radiographic assessment, Oxford Knee Score, SF12 and survivorship analysis. | Pre surgery, surgery, 3 month, 1, 3, 5 and 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Musgrave Park Hospital, Belfast, Ireland